CLINICAL TRIAL: NCT05319756
Title: A Phase 4 Randomized Double-blind Double-dummy Placebo & Active-controlled Single-dose Six-way Crossover Study Evaluating Abuse Potential of NEURONTIN® Taken Orally With Oxycodone HCL in Healthy Non-drug Dependent Recreational Opioid Users
Brief Title: Study Evaluating the Abuse Potential of NEURONTIN® in Healthy Non-drug Dependent, Recreational Opioid Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Viatris Specialty LLC (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: A9451180
Record Dates: First submitted 2022-03-08; First posted 2022-04-08 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Abuse Potential
Keywords: Neurontin; Oxycodone; Abuse Liability; Gabapentin
MeSH Terms: interventions — Gabapentin; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- gabapentin 600 mg single dose (Experimental)
  Interventions: Drug: gabapentin 600 mg
- gabapentin 1200 mg single dose (Experimental)
  Interventions: Drug: gabapentin 1200 mg
- gabapentin 600 mg and oxycodone HCl 20 mg (Experimental)
  Interventions: Drug: gabapentin 600 mg and oxycodone HCl 20 mg
- gabapentin 1200 mg and oxycodone HCl 20 mg (Experimental)
  Interventions: Drug: gabapentin 1200 mg and oxycodone HCl 20 mg
- oxycodone HCl 20 mg single dose (Active Comparator)
  Interventions: Drug: oxycodone HCl 20 mg
- placebo single dose (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: gabapentin 600 mg — Participants will receive a single oral dose of gabapentin 600 mg and a placebo that looks like oxycodone HCl
  Arms: gabapentin 600 mg single dose
Drug: gabapentin 1200 mg — Participants will receive a single oral dose of gabapentin 1200 mg and a placebo that looks like oxycodone HCl
  Arms: gabapentin 1200 mg single dose
Drug: gabapentin 600 mg and oxycodone HCl 20 mg — Participants will receive a single oral dose of gabapentin 600 mg and oxycodone HCl 20 mg
  Arms: gabapentin 600 mg and oxycodone HCl 20 mg
Drug: gabapentin 1200 mg and oxycodone HCl 20 mg — Participants will receive a single oral dose of gabapentin 1200 mg and oxycodone HCl 20 mg
  Arms: gabapentin 1200 mg and oxycodone HCl 20 mg
Drug: oxycodone HCl 20 mg — Participants will receive a single oral dose of oxycodone HCl 20 mg and a placebo that looks like gabapentin
  Arms: oxycodone HCl 20 mg single dose
Drug: placebo — Participants will receive a single oral dose of a placebo that looks like gabapentin and a placebo that looks like oxycodone HCl
  Arms: placebo single dose

SUMMARY:
This will be a randomized, double-blind, double-dummy, placebo- and active-controlled, 6 treatment, 6-period crossover single-dose, Williams square design study in healthy male and/or female adult, non-drug-dependent recreational opioid users.

DETAILED DESCRIPTION:
The study includes Screening, a Qualification Phase consisting of a Naloxone Challenge and Drug Discrimination crossover study, a Treatment Phase and Follow-up. Following successful completion of the Qualification Phase the participants will be enrolled in the Treatment phase. The Treatment Phase is a randomized, double-blind, double dummy, placebo- and active controlled, 6 treatment, 10-sequence, 6 period crossover, single-dose, Williams square design study in healthy male and/or female adult, non drug-dependent recreational users. On Day 1 of each of the Treatment Phase 6 periods, which will be separated by a washout of at least 14 days, participants will receive an oral dose of either gabapentin 600 mg or 1200 mg alone, or concomitantly with a 20 mg dose of oxycodone HCl or 20 mg monotherapy of oxycodone HCl or a placebo. Study treatments will be administered under fasted conditions (overnight fast and no food until 4 hours after dosing). Water will be allowed without restriction until 1 hour prior to dosing and 1 hour after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of screening. Participants must meet reproductive criteria as outlined in the protocol.
2. Male and female participants who are overtly healthy. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination, vital signs, 12-lead ECG, and/or clinical laboratory tests.
3. Participants must have drug abuse experience with opioids; ie, must have used opioids for non-therapeutic purposes (ie, for psychoactive effects) on at least 10 occasions within the last year and at least once in the 8 weeks before the Screening Visit (Visit 1).
4. Participants must satisfactorily complete both the Naloxone Challenge and the Drug Discrimination.
5. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
6. Body mass index (BMI) of 17.5 to 34 kg/m2, inclusive; and a total body weight ≥50 kg (110 lb).
7. Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

1. Current or past diagnosis of any type of drug dependence within the past year. Diagnosis of substance and/or alcohol dependence (excluding caffeine and nicotine) will be assessed by the Investigator using the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria performed at Screening. Current drug use will be allowed if the candidate can produce a negative urine sample and are free of any signs/symptoms of withdrawal. The candidate will be informed if they have a positive breathalyzer test.
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
3. Any condition possibly affecting drug absorption (eg, gastrectomy) excluding cholecystectomy within 1 year prior to study.
4. Abnormal baseline EtCO2 <35mm Hg or >45 mm Hg.
5. Clinical or laboratory evidence of active hepatitis A infection or a history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C, and/or positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb).
6. Participants with active suicidal ideation or suicidal behavior within 5 years prior to Screening as determined through the use of the Columbia Suicide Severity Rating Scale (C-SSRS) or active ideation identified at Screening or on Day 0.
7. Participants with any history of sleep apnea, myasthenia gravis or glaucoma.
8. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
9. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. (Refer to Section 6.5 for additional details).
10. Herbal supplements, herbal medications and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of study medication.
11. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives (whichever is longer) preceding the first dose of investigational product used in this study.
12. Positive urine drug screen (UDS) for substances of abuse at each admission in Qualification and Treatment Phase, excluding tetrahydrocannabinol (THC). If a participant presents with a positive UDS excluding THC at any admission or any visit, the investigator, at his/her discretion, may reschedule a repeat of UDS until the UDS is negative, excluding THC, before the participate is permitted to participate in any phase of the study.
13. Unable to abstain from using THC during the Qualification and Treatment Phase of the study.
14. Has participated in, is currently participating in, or is seeking treatment for substance and/or alcohol related disorders (excluding nicotine and caffeine).
15. Has a positive alcohol breathalyzer or urine test at each admission to the study center during Qualification and Treatment Phases. Positive results may be repeated and/or participants re scheduled at the Investigator's discretions.
16. Participants are heavy smokers or users of other types of nicotine products (>20 cigarettes equivalents per day).
17. Participants are unable to abstain from smoking for at least 2 hours before and at least 8 hours after study drug administration.
18. Screening sitting blood pressure (BP) >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility. Repeated BP tests should be spaced at least 5 minutes apart.
19. Baseline (screening) 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval as determined by the Fridericia method (QTcF) >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
20. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >=1.5 × upper limit of normal (ULN);
    * Total bilirubin level >=1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN.
21. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
22. History of sensitivity to heparin or heparin induced thrombocytopenia.
23. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
24. History of hypersensitivity to gabapentin or oxycodone or any of the components in the formulation of the study products.
25. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Sponsor employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dik WH NG, PhD, Study Director — Viatris Inc.
Locations (1):
- Hassman Research Institute, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were entered into a Qualification phase involving a naloxone challenge test (to exclude subjects who were opioid dependent) and a drug discrimination test (to confirm they can tell the difference between oxycodone and placebo). Only subjects who passed the tests in the Qualification phase were randomized into the Treatment phase where they received the 6 different single dose study treatments, each separated by a washout of at least 4 days, in the order specified for Sequences 1-6 below
Groups:
- Sequence 1: Period 1: Oxycodone 20 mg; Period 2: Placebo; Period 3: Gabapentin 1200 mg plus Oxycodone 20 mg; Period 4: Gabapentin 600 mg; Period 5: Gabapentin 600 mg plus Oxycodone 20 mg; Period 6: Gabapentin 1200 mg
- Sequence 2: Period 1: Placebo; Period 2: Gabapentin 600 mg; Period 3: Oxycodone 20 mg; Period 4: Gabapentin 1200 mg; Period 5: Gabapentin 1200 mg plus Oxycodone 20 mg; Period 6: Gabapentin 600 mg plus Oxycodone 20 mg
- Sequence 3: Period 1: Gabapentin 600 mg; Period 2: Gabapentin 1200 mg; Period 3: Placebo; Period 4 Gabapentin 600 mg plus Oxycodone 20 mg; Period 5: Oxycodone 20 mg; Period 6: Gabapentin 1200 mg plus Oxycodone 20 mg
- Sequence 4: Period 1: Gabapentin 1200 mg; Period 2: Gabapentin 600 mg plus Oxycodone 20 mg; Period 3: Gabapentin 600 mg; Period 4: Gabapentin 1200 mg plus Oxycodone 20 mg; Period 5: Placebo; Period 6: Oxycodone 20 mg
- Sequence 5: Period 1: Gabapentin 600 mg plus Oxycodone 20 mg; Period 2: Gabapentin 1200 mg plus Oxycodone 20 mg; Period 3: Gabapentin 1200 mg; Period 4: Oxycodone 20 mg; Period 5: Gabapentin 600 mg; Period 6: Placebo
- Sequence 6: Period 1: Gabapentin 1200 mg plus Oxycodone 20 mg; Period 2: Oxycodone 20 mg; Period 3: Gabapentin 600 mg plus Oxycodone 20 mg; Period 4: Placebo; Period 5: Gabapentin 1200 mg; Period 6: Gabapentin 600 mg
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed | 8 | 8 | 9 | 9 | 8 | 8
Not Completed | 1 | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants who were randomized to a treatment sequence in the Treatment Phase.
Groups:
- Randomized Population: All participants who were randomized to a treatment sequence in the Treatment Phase.
Arm/Group | Randomized Population
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 35
  White | 13
  More than one race | 4
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Bipolar Visual Analog Scale (VAS) for "Drug Liking" Maximum Effect (Emax).
Description: Drug liking assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: up to 48 hours after treatments
Population: The analysis population was the modified completer population which included subjects who completed all 6 treatment periods but excluded those identified during data review as having maximum Drug Liking scores that were similar for all 6 treatments or who had high placebo responses
Measure: Mean (Standard Error); unit: Score on a 100 mm scale
Groups:
- Placebo: Participants received a single oral dose of a placebo that looks like gabapentin and a placebo that looks like oxycodone HCl
- Oxycodone HCl 20 mg Single Dose: Participants received a single oral dose of oxycodone HCl 20 mg and a placebo that looks like gabapentin
- Gabapentin 600 mg Single Dose: Participants received a single oral dose of gabapentin 600 mg and a placebo that looks like oxycodone HCl
- Gabapentin 1200 mg Single Dose: Participants received a single oral dose of gabapentin 1200 mg and a placebo that looks like oxycodone HCl
- Gabapentin 600 mg and Oxycodone HCl 20 mg: Participants received a single oral dose of gabapentin 600 mg and oxycodone HCl 20 mg
- Gabapentin 1200 mg and Oxycodone HCl 20 mg: Participants received a single oral dose of gabapentin 1200 mg and oxycodone HCl 20 mg
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
Score on a 100 mm scale | 54.89 (2.116) | 87.40 (3.156) | 57.89 (3.142) | 63.62 (3.334) | 88.43 (3.216) | 92.17 (2.713)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone HCl 20 mg Single Dose; The sensitivity and integrity of the study was validated by comparing the mean responses of oxycodone HCl, the positive control (C), to the placebo (P): H0: μC - μP ≤ δ1 versus Ha: μC - μP > δ1 where δ1 =15; Test type: Superiority; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 32.8, 95% CI 1-sided [lower limit 26.1], Standard Error of Mean 4.00
Statistical Analysis 2: Comparison: Placebo vs Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; The primary analysis evaluated whether gabapentin plus oxycodone HCl (T) produced mean responses that showed abuse potential that was no higher than oxycodone HCl (C). The margin for showing no significant difference was defined as 20% of the difference between oxycodone HCl (C) and Placebo (P): H0: μT - μC ≥ 0.2(μC - μP) versus Ha: μT - μC <0.2(μC - μP); Test type: Non-Inferiority — Non-inferiority margin = 0; p = 0.1041, Mixed Models Analysis; Mean Difference (Final Values) = -5.6, 95% CI 1-sided [upper limit 1.7], Standard Error of Mean 4.46
Statistical Analysis 3: Comparison: Placebo vs Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority margin = 0; p = 0.3373, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 1-sided [upper limit 5.5], Standard Error of Mean 4.46
Statistical Analysis 4: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; The null and alternative hypotheses for evaluating whether gabapentin (G) produced mean responses that show less abuse potential than oxycodone HCl (C) were: H0: μC - μG ≤ 0.2(μC - 50) versus Ha: μC - μG >0.2(μC - 50); Test type: Non-Inferiority — Non-inferiority margin = 10; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -12.3, 95% CI 1-sided [upper limit -6.3], Standard Error of Mean 3.63
Statistical Analysis 5: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority — Non-inferiority margin = 10; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -6.7, 95% CI 1-sided [upper limit -0.6], Standard Error of Mean 3.64
Statistical Analysis 6: Comparison: Placebo vs Gabapentin 600 mg Single Dose; The null and alternative hypotheses for evaluating whether gabapentin (G) produced mean responses that show abuse potential similar to placebo(P) were: H0: μG - μP ≥ δ2 versus Ha: μG - μP < δ2 where δ2 =11; Test type: Non-Inferiority — Non-inferiority margin = 11; p = 0.0232, Mixed Models Analysis; Mean Difference (Final Values) = 3.0, 95% CI 1-sided [upper limit 9.6], Standard Error of Mean 4.00
Statistical Analysis 7: Comparison: Placebo vs Gabapentin 1200 mg Single Dose; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority — Non-inferiority margin = 11; p = 0.2767, Mixed Models Analysis; Mean Difference (Final Values) = 8.6, 95% CI 1-sided [upper limit 15.2], Standard Error of Mean 4.01

2. Secondary Outcome: Bipolar VAS for "Drug Liking" - Time to Maximum Effect (TEmax)
Description: Time after dosing when the maximum effect for Drug Liking VAS is reached
Time Frame: up to 48 hours after treatments
Population: Modified completer population
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Single Dose | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
hours | 0.25 [0.2 to 24.0] | 1.00 [0.2 to 3.5] | 0.25 [0.25 to 2.5] | 0.28 [0.1 to 12.1] | 1.00 [0.2 to 12.0] | 1.50 [0.2 to 4.0]

3. Secondary Outcome: Bipolar VAS for "Drug Liking": Area Under the Effect Curve From Time 0 to the Last Available Data (AUEClast)
Description: Area under the effect-time profile from time 0 to the time of the last available data for the "Drug liking" visual analog scale which assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: Up to 48 hours after treatments (Assessments were made at the following timepoints after each treatment: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, and 48 hours)
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Groups:
- Placebo Single Dose: Participants will receive a single oral dose of a placebo that looks like gabapentin and a placebo that looks like oxycodone HCl
- Oxycodone HCl 20 mg Single Dose: Participants will receive a single oral dose of oxycodone HCl 20 mg and a placebo that looks like gabapentin
- Gabapentin 600 mg Single Dose: Participants will receive a single oral dose of gabapentin 600 mg and a placebo that looks like oxycodone HCl
- Gabapentin 1200 mg Single Dose: Participants will receive a single oral dose of gabapentin 1200 mg and a placebo that looks like oxycodone HCl
Arm/Group | Placebo Single Dose | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
units on a scale * hour | 2394.21 (65.274) | 2661.43 (84.274) | 2422.37 (85.855) | 2444.4 (83.580) | 2744.86 (76.342) | 2759.57 (74.589)
Statistical Analysis 1: Comparison: Placebo Single Dose vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = 267.1, 90% CI 2-sided [128.8 to 405.4], Standard Error of Mean 83.688
Statistical Analysis 2: Comparison: Placebo Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.7276, Mixed Models Analysis; Mean Difference (Final Values) = 29.19, 90% CI 2-sided [-109 to 167.5], Standard Error of Mean 83.688
Statistical Analysis 3: Comparison: Placebo Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.5481, Mixed Models Analysis; Mean Difference (Final Values) = 50.41, 90% CI 2-sided [-88.0 to 188.9], Standard Error of Mean 83.785
Statistical Analysis 4: Comparison: Placebo Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 350.7, 90% CI 2-sided [211.8 to 489.5], Standard Error of Mean 84.023
Statistical Analysis 5: Comparison: Placebo Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 364.4, 90% CI 2-sided [225.9 to 502.8], Standard Error of Mean 83.785
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.0050, Mixed Models Analysis; Mean Difference (Final Values) = -238, 90% CI 2-sided [-376 to -99.4], Standard Error of Mean 83.785
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.0106, Mixed Models Analysis; Mean Difference (Final Values) = -217, 90% CI 2-sided [-356 to -77.8], Standard Error of Mean 84.023
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.3196, Mixed Models Analysis; Mean Difference (Final Values) = 83.60, 90% CI 2-sided [-54.9 to 222.1], Standard Error of Mean 83.785
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.2464, Mixed Models Analysis; Mean Difference (Final Values) = 97.29, 90% CI 2-sided [-41.0 to 235.6], Standard Error of Mean 83.688

4. Secondary Outcome: Bipolar VAS for "Drug Liking": Area Under the Effect Curve to 1 Hour (AUEC1)
Description: Area under the effect-time profile from time 0 to 1 hour post-dose for the "Drug liking" visual analog scale which assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: Up to 1 hour post-dose (Assessments were made at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, and 1 hour)
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
units on a scale * hour | 50.17 (0.317) | 58.86 (1.478) | 51.28 (1.440) | 50.61 (0.568) | 57.02 (1.771) | 55.76 (1.390)

5. Secondary Outcome: Bipolar VAS for "Drug Liking": Area Under the Effect Curve to 2 Hours (AUEC2)
Description: Area under the effect-time profile from time 0 to 2 hours post-dose for the "Drug liking" visual analog scale which assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: Up to 2 hours after treatments (Assessments were made at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, 1, 1.5, and 2 hours)
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
units on a scale * hour | 102.62 (1.791) | 140.44 (4.434) | 105.20 (4.017) | 107.19 (2.449) | 138.72 (4.340) | 133.84 (4.010)

6. Secondary Outcome: Bipolar VAS for "Drug Liking": Area Under the Effect Curve to 3 Hours (AUEC3)
Description: Area under the effect-time profile from time 0 to 3 hours post-dose for the "Drug liking" visual analog scale which assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: up to 3 hours after treatments (Assessments were made at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, and 3 hours)
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
units on a scale * hour | 155.48 (3.651) | 219.31 (7.614) | 161.07 (6.535) | 164.03 (4.819) | 223.22 (7.326) | 214.99 (6.567)

7. Secondary Outcome: Bipolar VAS for "Drug Liking": Area Under the Effect Curve to 4 Hours (AUEC4)
Description: Area under the effect-time profile from time 0 to 4 hours post-dose for the "Drug liking" visual analog scale which assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: Up to 4 hours after treatments (Assessments were made at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, and 4 hours)
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
units on a scale * hour | 208.32 (5.171) | 294.28 (10.329) | 214.53 (8.878) | 220.08 (6.896) | 305.08 (10.423) | 293.99 (8.810)

8. Secondary Outcome: Bipolar VAS for "Drug Liking": Area Under the Effect Curve to 8 Hours (AUEC8)
Description: Area under the effect-time profile from time 0 to 8 hours post-dose for the "Drug liking" visual analog scale which assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: Up to 8 hours after treatments (Assessments were made at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours)
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
units on a scale * hour | 411.58 (12.224) | 551.53 (19.517) | 421.12 (17.144) | 438.30 (13.862) | 599.96 (22.312) | 574.98 (18.952)

9. Secondary Outcome: Unipolar VAS for "High" - Maximum Effect (Emax)
Description: Maximum effect on the 100 mm visual analog scale for the question "I am feeling high" where 0 = "not at all" and 100 = "extremely"
Time Frame: up to 48 hours after treatments
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo Single Dose | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
Score on a 100 mm scale | 13.45 (4.854) | 77.36 (5.8160) | 28.61 (6.551) | 25.21 (6.412) | 81.86 (5.620) | 88.74 (4.210)
Statistical Analysis 1: Comparison: Placebo Single Dose vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 64.67, 90% CI 2-sided [52.15 to 77.20], Standard Error of Mean 7.581
Statistical Analysis 2: Comparison: Placebo Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.0546, Mixed Models Analysis; Mean Difference (Final Values) = 14.66, 90% CI 2-sided [2.13 to 27.1], Standard Error of Mean 7.581
Statistical Analysis 3: Comparison: Placebo Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.1286, Mixed Models Analysis; Mean Difference (Final Values) = 11.58, 90% CI 2-sided [-0.96 to 24.12], Standard Error of Mean 7.589
Statistical Analysis 4: Comparison: Placebo Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 68.99, 90% CI 2-sided [56.42 to 81.57], Standard Error of Mean 7.611
Statistical Analysis 5: Comparison: Placebo Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 76.37, 90% CI 2-sided [63.83 to 88.91], Standard Error of Mean 7.589
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -50.0, 90% CI 2-sided [-62.6 to -37.5], Standard Error of Mean 7.589
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -53.1, 90% CI 2-sided [-65.7 to -40.5], Standard Error of Mean 7.611
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.5699, Mixed Models Analysis; Mean Difference (Final Values) = 4.32, 90% CI 2-sided [-8.22 to 16.86], Standard Error of Mean 7.589
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.1243, Mixed Models Analysis; Mean Difference (Final Values) = 11.70, 90% CI 2-sided [-0.83 to 24.23], Standard Error of Mean 7.581

10. Secondary Outcome: Unipolar VAS for "High": Time to Maximum Effect (TEmax)
Description: Time after dosing when the maximum effect for "High" VAS is reached
Time Frame: up to 48 hours after treatments
Population: Modified completer population
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Single Dose | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
hours | 0.25 [0.2 to 8.0] | 1.00 [0.3 to 4.0] | 0.26 [0.2 to 8.0] | 0.27 [0.1 to 144.9] | 1.00 [0.2 to 48.1] | 1.50 [0.2 to 4.1]

11. Secondary Outcome: Area Under the Effect Curve for "High" VAS (AUEClast)
Description: Area under the effect-time profile from time 0 to the time of the last available data for the "High" visual analog scale which measures on a 100 mm visual analog scale the subject's response to the question "I am feeling high" where 0 = "not at all" and 100 ="extremely"
Time Frame: as for outcome 3
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo Single Dose | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
units on a scale * hour | 33.45 (14.904) | 321.75 (46.346) | 86.41 (31.541) | 123.74 (50.060) | 512.08 (66.299) | 425.01 (52.651)
Statistical Analysis 1: Comparison: Placebo Single Dose vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 286.7, 90% CI 2-sided [202.6 to 370.8], Standard Error of Mean 50.879
Statistical Analysis 2: Comparison: Placebo Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.2912, Mixed Models Analysis; Mean Difference (Final Values) = 53.85, 90% CI 2-sided [-30.2 to 137.9], Standard Error of Mean 50.879
Statistical Analysis 3: Comparison: Placebo Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.0563, Mixed Models Analysis; Mean Difference (Final Values) = 97.80, 90% CI 2-sided [13.62 to 182.0], Standard Error of Mean 50.938
Statistical Analysis 4: Comparison: Placebo Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 484.5, 90% CI 2-sided [400.1 to 569.0], Standard Error of Mean 51.083
Statistical Analysis 5: Comparison: Placebo Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 396.6, 90% CI 2-sided [312.4 to 480.8], Standard Error of Mean 50.938
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -233, 90% CI 2-sided [-317 to -149], Standard Error of Mean 50.938
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -189, 90% CI 2-sided [-273 to -105], Standard Error of Mean 51.083
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 197.8, 90% CI 2-sided [113.7 to 282.0], Standard Error of Mean 50.938
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0320, Mixed Models Analysis; Mean Difference (Final Values) = 109.9, 90% CI 2-sided [25.80 to 194.0], Standard Error of Mean 50.879

12. Secondary Outcome: Bipolar VAS for "Take Drug Again"
Description: 100 mm visual analog scale at 24, 36, and 48 hours post-dose for the question "I would take this drug again" where 0 = "definitely not", 50 = "neutral", and 100 = "definitely so". The data from the 24, 36, and 48 hours postdose measurements were combined into a single overall model-adjusted value for 24 to 48 hours post-treatment timeframe by estimation from a mixed model with treatment, period, treatment sequence, time, and treatment*time as fixed effects, subject nested within sequence as a random effect. The compound symmetric covariance matrix was employed. Data from all time points were included
Time Frame: Up to 48 hours after treatments (Assessments were made at the following timepoints after each treatment for this outcome measure: 24, 36, and 48 hours)
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo Single Dose | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
Score on a 100 mm scale | 53.43 (2.928) | 72.16 (2.918) | 55.19 (2.942) | 58.05 (2.935) | 79.16 (2.940) | 77.85 (2.910)
Statistical Analysis 1: Comparison: Placebo Single Dose vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 18.73, 90% CI 2-sided [14.98 to 22.48], Standard Error of Mean 2.276
Statistical Analysis 2: Comparison: Placebo Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.5056, Mixed Models Analysis; Mean Difference (Final Values) = 1.76, 90% CI 2-sided [-2.03 to 5.56], Standard Error of Mean 2.302
Statistical Analysis 3: Comparison: Placebo Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.0760, Mixed Models Analysis; Mean Difference (Final Values) = 4.62, 90% CI 2-sided [0.82 to 8.42], Standard Error of Mean 2.307
Statistical Analysis 4: Comparison: Placebo Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 25.73, 90% CI 2-sided [21.92 to 29.54], Standard Error of Mean 2.315
Statistical Analysis 5: Comparison: Placebo Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 24.42, 90% CI 2-sided [20.68 to 28.16], Standard Error of Mean 2.270
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -17.0, 90% CI 2-sided [-20.8 to -13.2], Standard Error of Mean 2.297
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -14.1, 90% CI 2-sided [-17.9 to -10.3], Standard Error of Mean 2.299
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0024, Mixed Models Analysis; Mean Difference (Final Values) = 7.00, 90% CI 2-sided [3.22 to 10.79], Standard Error of Mean 2.298
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0118, Mixed Models Analysis; Mean Difference (Final Values) = 5.69, 90% CI 2-sided [1.98 to 9.41], Standard Error of Mean 2.255

13. Secondary Outcome: Bipolar VAS for "Overall Drug Liking"
Description: 100 mm visual analog scale at 24, 36, and 48 hours post-dose for the question "Overall, my liking for this drug is" where 0 = "definitely not", 50 = "neutral", and 100 = "definitely so". The data from the 24, 36, and 48 hours postdose measurements were combined into a single overall model-adjusted value for 24 to 48 hours post-treatment timeframe by estimation from a mixed model with treatment, period, treatment sequence, time, and treatment*time as fixed effects, subject nested within sequence as a random effect. The compound symmetric covariance matrix was employed. Data from all time points were included
Time Frame: as for outcome 12
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo Single Dose | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
Score on a 100 mm scale | 51.75 (2.895) | 72.06 (2.886) | 54.40 (2.909) | 58.25 (2.902) | 75.90 (2.907) | 79.94 (2.878)
Statistical Analysis 1: Comparison: Placebo Single Dose vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 20.31, 90% CI 2-sided [16.61 to 24.01], Standard Error of Mean 2.246
Statistical Analysis 2: Comparison: Placebo Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.2439, Mixed Models Analysis; Mean Difference (Final Values) = 2.65, 90% CI 2-sided [-1.09 to 6.39], Standard Error of Mean 2.271
Statistical Analysis 3: Comparison: Placebo Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.0044, Mixed Models Analysis; Mean Difference (Final Values) = 6.50, 90% CI 2-sided [2.75 to 10.25], Standard Error of Mean 2.276
Statistical Analysis 4: Comparison: Placebo Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 24.15, 90% CI 2-sided [20.39 to 27.91], Standard Error of Mean 2.284
Statistical Analysis 5: Comparison: Placebo Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 28.19, 90% CI 2-sided [24.50 to 31.88], Standard Error of Mean 2.240
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -17.7, 90% CI 2-sided [-21.4 to -13.9], Standard Error of Mean 2.266
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -13.8, 90% CI 2-sided [-17.5 to -10.1], Standard Error of Mean 2.268
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0907, Mixed Models Analysis; Mean Difference (Final Values) = 3.84, 90% CI 2-sided [0.11 to 7.57], Standard Error of Mean 2.267
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 7.88, 90% CI 2-sided [4.22 to 11.55], Standard Error of Mean 2.225

14. Secondary Outcome: Unipolar VAS for "Good Drug Effect"
Description: 100 mm visual analog scale for the question "At this moment, I can feel good drug effects" where 0 = "not at all" and 100 = "extremely"
Time Frame: up to 48 hours after treatments
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
Score on a 100 mm scale | 2.54 (2.123) | 27.91 (2.117) | 6.13 (2.117) | 8.73 (2.120) | 34.72 (2.119) | 32.71 (2.113)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 25.37, 90% CI 2-sided [22.86 to 27.88], Standard Error of Mean 1.528
Statistical Analysis 2: Comparison: Placebo vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.0189, Mixed Models Analysis; Mean Difference (Final Values) = 3.59, 90% CI 2-sided [1.08 to 6.11], Standard Error of Mean 1.529
Statistical Analysis 3: Comparison: Placebo vs Gabapentin 1200 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.18, 90% CI 2-sided [3.66 to 8.71], Standard Error of Mean 1.536
Statistical Analysis 4: Comparison: Placebo vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 32.18, 90% CI 2-sided [29.65 to 34.71], Standard Error of Mean 1.537
Statistical Analysis 5: Comparison: Placebo vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 30.17, 90% CI 2-sided [27.66 to 32.68], Standard Error of Mean 1.525
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -21.8, 90% CI 2-sided [-24.3 to -19.3], Standard Error of Mean 1.522
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -19.2, 90% CI 2-sided [-21.7 to -16.7], Standard Error of Mean 1.530
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.81, 90% CI 2-sided [4.30 to 9.31], Standard Error of Mean 1.524
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = 4.80, 90% CI 2-sided [2.31 to 7.29], Standard Error of Mean 1.514

15. Secondary Outcome: Unipolar VAS for "Bad Drug Effect"
Description: 100 mm visual analog scale for the question "At this moment, I can feel bad drug effects" where 0 = "not at all" and 100 = "extremely"
Time Frame: up to 48 hours after treatments
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
Score on a 100 mm scale | 0.19 (1.211) | 4.41 (1.209) | 0.82 (1.209) | 0.97 (1.210) | 4.10 (1.210) | 3.41 (1.207)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.23, 90% CI 2-sided [3.01 to 5.45], Standard Error of Mean 0.743
Statistical Analysis 2: Comparison: Placebo vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.3933, Mixed Models Analysis; Mean Difference (Final Values) = 0.63, 90% CI 2-sided [-0.59 to 1.86], Standard Error of Mean 0.743
Statistical Analysis 3: Comparison: Placebo vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.2916, Mixed Models Analysis; Mean Difference (Final Values) = 0.79, 90% CI 2-sided [-0.44 to 2.02], Standard Error of Mean 0.747
Statistical Analysis 4: Comparison: Placebo vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.92, 90% CI 2-sided [2.69 to 5.15], Standard Error of Mean 0.748
Statistical Analysis 5: Comparison: Placebo vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.22, 90% CI 2-sided [2.00 to 4.44], Standard Error of Mean 0.742
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.59, 90% CI 2-sided [-4.81 to -2.38], Standard Error of Mean 0.740
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.44, 90% CI 2-sided [-4.66 to -2.22], Standard Error of Mean 0.744
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.6765, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 90% CI 2-sided [-1.53 to 0.91], Standard Error of Mean 0.741
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.1712, Mixed Models Analysis; Mean Difference (Final Values) = -1.01, 90% CI 2-sided [-2.22 to 0.20], Standard Error of Mean 0.737

16. Secondary Outcome: Unipolar VAS for "Any Drug Effect"
Description: 100 mm visual analog scale for the question "At this moment, I can feel any drug effects" where 0 = "not at all" and 100 = "extremely"
Time Frame: up to 48 hours after treatments
Population: Modified completer population
Measure: Least Squares Mean (Standard Error); unit: Score on a 100 mm scale
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42
Score on a 100 mm scale | 3.77 (2.167) | 28.46 (2.161) | 6.63 (2.162) | 7.88 (2.164) | 34.34 (2.163) | 33.76 (2.158)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone HCl 20 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 24.70, 90% CI 2-sided [22.19 to 27.21], Standard Error of Mean 1.526
Statistical Analysis 2: Comparison: Placebo vs Gabapentin 600 mg Single Dose; Test type: Other; p = 0.0606, Mixed Models Analysis; Mean Difference (Final Values) = 2.87, 90% CI 2-sided [0.35 to 5.38], Standard Error of Mean 1.527
Statistical Analysis 3: Comparison: Placebo vs Gabapentin 1200 mg Single Dose; Test type: Other; p = 0.0074, Mixed Models Analysis; Mean Difference (Final Values) = 4.11, 90% CI 2-sided [1.59 to 6.64], Standard Error of Mean 1.534
Statistical Analysis 4: Comparison: Placebo vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 30.58, 90% CI 2-sided [28.05 to 33.10], Standard Error of Mean 1.536
Statistical Analysis 5: Comparison: Placebo vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 29.99, 90% CI 2-sided [27.48 to 32.50], Standard Error of Mean 1.524
Statistical Analysis 6: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -21.8, 90% CI 2-sided [-24.3 to -19.3], Standard Error of Mean 1.521
Statistical Analysis 7: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg Single Dose; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -20.6, 90% CI 2-sided [-23.1 to -18.1], Standard Error of Mean 1.529
Statistical Analysis 8: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 600 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.88, 90% CI 2-sided [3.37 to 8.38], Standard Error of Mean 1.523
Statistical Analysis 9: Comparison: Oxycodone HCl 20 mg Single Dose vs Gabapentin 1200 mg and Oxycodone HCl 20 mg; Test type: Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = 5.29, 90% CI 2-sided [2.80 to 7.78], Standard Error of Mean 1.513

17. Secondary Outcome: Cmax of Gabapentin
Description: Maximum plasma concentration of gabapentin
Time Frame: Up to 48 hours after treatments (concentrations were measured at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, and 48 hours)
Population: Pharmacokinetic population: all enrolled participants who received study medication and have pharmacokinetic data for the parameters of interest.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 52 | 52 | 52
micrograms/milliliter | 4.16 (1.422) | 6.07 (1.951) | 4.17 (1.121) | 6.18 (1.443)

18. Secondary Outcome: Tmax of Gabapentin
Description: Time when the maximum concentration of gabapentin is reached
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: Hours
Arm/Group | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 52 | 52 | 52
Hours | 3.13 [1.2 to 6.1] | 3.13 [1.6 to 6.1] | 3.13 [1.2 to 8.1] | 3.13 [1.2 to 8.2]

19. Secondary Outcome: AUCinf of Gabapentin
Description: Area under the plasma concentration/time curve from time 0 extrapolated to infinity time of gabapentin
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter
Arm/Group | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 52 | 52 | 52
micrograms*hour/milliliter | 41.42 (11.798) | 65.38 (18.854) | 48.58 (12.009) | 75.18 (18.431)

20. Secondary Outcome: AUClast of Gabapentin
Description: Area under the plasma concentration/time profile from time 0 to the time of the last quantifiable concentration of gabapentin
Time Frame: Up to 48 hours after treatment (concentrations were measured at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, and 48 hours)
Population: Pharmacokinetic population: all enrolled participants who received study medication and have pharmacokinetic data for the parameters of interes
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter
Arm/Group | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 52 | 52 | 52
micrograms*hour/milliliter | 39.76 (11.856) | 61.42 (19.900) | 47.31 (12.142) | 72.73 (17.781)

21. Secondary Outcome: Half-life (t½) of Gabapentin
Description: Half-life (t½) of gabapentin
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 51 | 52 | 52
Hours | 9.14 (10.846) | 10.62 (7.674) | 8.20 (3.551) | 9.19 (3.596)

22. Secondary Outcome: Cmax of Oxycodone
Description: Maximum plasma concentration of Oxycodone
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 51 | 50
nanograms/milliliter | 44.92 (17.336) | 43.82 (14.144) | 40.79 (14.809)

23. Secondary Outcome: Tmax of Oxycodone
Description: Time when the maximum concentration of Oxycodone is reached
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 51 | 50
hours | 1.15 [0.6 to 8.1] | 1.15 [0.6 to 5.9] | 1.63 [0.6 to 3.6]

24. Secondary Outcome: AUCinf of Oxycodone
Description: Area under the plasma concentration/time curve from time 0 extrapolated to infinity time of Oxycodone
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter
Arm/Group | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 51 | 49
nanograms*hour/milliliter | 233.29 (64.369) | 228.40 (71.854) | 234.94 (77.115)

25. Secondary Outcome: AUClast of Oxycodone
Description: Area under the plasma concentration/time profile from time 0 to the time of the last quantifiable concentration of Oxycodone
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter
Arm/Group | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 51 | 50
nanograms*hour/milliliter | 229.31 (64.935) | 224.79 (71.748) | 234.65 (80.068)

26. Secondary Outcome: Half-life (t½) of Oxycodone
Description: Half-life (t½) of Oxycodone
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
Number analyzed (Participants) | 51 | 51 | 49
hours | 4.12 [2.6 to 6.2] | 3.84 [2.2 to 6.1] | 3.90 [2.4 to 10.7]

ADVERSE EVENTS:
Time Frame: During the entire Treatment Phase of the study, which encompassed the time interval from admission of the subject to their first Treatment Period until 28 days after study drug dosing in their last (6th) Treatment Period, including the washout in between Treatment Periods. The total duration of the Treatment Phase for each subject was dependent on visit scheduling and whether the subject completed all 6 treatment periods, and it lasted up to approximately 13 weeks.
Description: Adverse events that occur during the washout interval between treatment visits or during the follow up after the final study drug dose were counted under the previous treatment visit
Arm/Group | Placebo | Oxycodone HCl 20 mg Single Dose | Gabapentin 600 mg Single Dose | Gabapentin 1200 mg Single Dose | Gabapentin 600 mg and Oxycodone HCl 20 mg | Gabapentin 1200 mg and Oxycodone HCl 20 mg
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52 | 0/51 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/51 | 0/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 4/52 | 0/51 | 2/52 | 4/52 | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=53) | Oxycodone HCl 20 mg Single Dose (N=52) | Gabapentin 600 mg Single Dose (N=51) | Gabapentin 1200 mg Single Dose (N=52) | Gabapentin 600 mg and Oxycodone HCl 20 mg (N=52) | Gabapentin 1200 mg and Oxycodone HCl 20 mg (N=52)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT05319756/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT05319756/SAP_001.pdf